CLINICAL TRIAL: NCT01975142
Title: Validity of HER2-amplified Circulating Tumor Cells to Select Metastatic Breast Cancer Considered HER2-negative for Trastuzumab-emtansine (T-DM1) Treatment.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IC 2013-03
Record Dates: First submitted 2013-10-17; First posted 2013-11-04 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Breast Cancer, HER2 Negative Primary Tumor
Keywords: Metastatic breast cancer; HER2 negative primary tumor; CTC HER2 positive
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TDM-1 (Experimental)
  Interventions: Drug: Trastuzumab - Emtansine

INTERVENTIONS:
Drug: Trastuzumab - Emtansine

SUMMARY:
Patients with metastatic breast cancer considered HER2 negative are screened for HER2-amplified circulating tumor cells. If at least HER2-amplified circulating tumor cell is detected, patients are treated by Trastuzumab - Emtansine (T-DM1) in a single arm phase II with an adaptive design.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for screening:

* Breast adenocarcinoma considered HER2-negative on the primary tumour or unknown status HER2
* A least one metastatic site and/or inoperable loco-regional relapse
* Measurable disease (RECIST v1.1)
* Age from 18 to 75 years
* Performance status of 0-2
* Efficient contraceptive in non-menopause women

Inclusion criteria for treatment :

* At least 1 (Cohort " L ") or 3 (cohort " H ") HER2 amplified CTC
* Performance status of 0-2
* Adequate cardiac function
* Adequate hematological and biochemical blood tests

Exclusion Criteria:

* Life expectancy of less than 3 months
* Previous history of any other stage III or IV invasive cancer
* Male breast cancer
* Uncontrolled brain metastases
* Significant cumulated exposure to anthracyclines
* Current or previous significant history of cardio-vascular/pulmonary disease
* Previous use of trastuzumab

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2013-11-07 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2019-01-21 (Actual)

PRIMARY OUTCOMES:
Tumor response rate to T-DM1 in patients with HER2 amplified circulating tumor cells | Until disease progression (estimated duration : 1 year)
  Assessment every 6 weeks.

SECONDARY OUTCOMES:
Detection rate of HER2 amplified circulating tumor cells, heterogeneity rate between circulating tumor cells and correlations with patient characteristics | 1 month
Technical failure rate and reproducibility of HER2 FISH on circulating tumor cells | 1 month
Correlation between HER2 FISH and immunofluorescence on circulating tumor cells | 1 month
Progression-free survival | 4 years
Disease control rate (responses and stable diseases) | Until disease progression (estimated duration : 1 year)
Correlation between treatment efficacy and HER2 FISH results (level of amplification, absolute number and percentage of amplified cells) | Until disease progression (estimated duration : 1 year)
Changes in CTC numbers during treatment | Until disease progression (estimated duration : 1 year)
Circulating tumor DNA before and during treatment | Until disease progression (estimated duration : 1 year)
Treatment toxicity | Until disease progression (estimated duration : 1 year)
  Toxicity of the treatment from first intake until disease progression

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Clinique Victor Hugo, Le Mans
  - Institut de Cancérologie HARTMANN, Levallois-Perret
  - Centre Oscar Lambret, Lille
  - Chu de Limoges, Limoges
  - Centre Val d'Aurelle - P. Lamarque, Montpellier
  - Institut Curie, Paris
  - Chu Saint-Louis, Paris
  - Institut Curie - Hôpital René HUGENIN, Saint-Cloud
  - Centre Catherine de Sienne, Vandœuvre-lès-Nancy
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jacot W, Cottu P, Berger F, Dubot C, Venat-Bouvet L, Lortholary A, Bourgeois H, Bollet M, Servent V, Luporsi E, Espie M, Guiu S, D'Hondt V, Dieras V, Sablin MP, Brain E, Neffati S, Pierga JY, Bidard FC. Actionability of HER2-amplified circulating tumor cells in HER2-negative metastatic breast cancer: the CirCe T-DM1 trial. Breast Cancer Res. 2019 Nov 14;21(1):121. doi: 10.1186/s13058-019-1215-z. PMID 31727113